CLINICAL TRIAL: NCT05105516
Title: Diagnosis Of Early Cardiac Dysfunction in Patients With Idiopathic Frequent Monomorphic PVCs and Effect Effect of Ablation and Comparison Between Different Sites of Ablation
Brief Title: Diagnosis Of Early Cardiac Dysfunction in Patients With Idiopathic Frequent Monomorphic PVCs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Usama Mohammed Tony, MTony, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cardiomyopathy in PVCs
Record Dates: First submitted 2021-10-25; First posted 2021-11-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Cardiomyopathies
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ablation (Other): Comparison between different sites of ablation
  Interventions: Procedure: Ablation

INTERVENTIONS:
Procedure: Ablation — Ablation of ectopic foci causing PVCs

SUMMARY:
Diagnosis Of Early Cardiac Dysfunction in Patients With Idiopathic Frequent Monomorphic PVCs and effect of ablation and comparison between different sites of ablation

DETAILED DESCRIPTION:
* Apply the speckle myocardial tracking technology to early diagnose dysfunction in patients with idiopathic frequent monomorphic PVCs
* Assessment of cardiac function before and after ablation and comparison before and after ablation and between sites of origin of the PVCs as diagnosed by the electrophysiologic and 3d mapping techniques that may be more confirmed by successful ablation whenever achieved

ELIGIBILITY:
Inclusion Criteria:

* All patients of sample size admitted to the cardiology department of Assiut university hospital for ablation of idiopathic frequent monomorphic PVCs

Exclusion Criteria:

* Patients with well-known factors of cardiac dysfunctions, including high blood pressure (over 140/90 mmHg), hypertrophic cardiomyopathy, left ventricular hypertrophy, bundle branch block, severe valvular disease, complete heart block, and previous CABG.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
• Detection of early cardiac dysfunction in patients with idiopathic frequent monomorphic PVCs . | Baseline
  • Assessment of cardiac function in patients with idiopathic frequent monomorphic PVCs post - ablation and patients on medical treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Latchamsetty R, Bogun F. Premature Ventricular Complex-Induced Cardiomyopathy. JACC Clin Electrophysiol. 2019 May;5(5):537-550. doi: 10.1016/j.jacep.2019.03.013. PMID 31122375
- [Background] Sharma E, Arunachalam K, Di M, Chu A, Maan A. PVCs, PVC-Induced Cardiomyopathy, and the Role of Catheter Ablation. Crit Pathw Cardiol. 2017 Jun;16(2):76-80. doi: 10.1097/HPC.0000000000000106. PMID 28509708